CLINICAL TRIAL: NCT00214539
Title: Multicenter Randomized Clinical Trial of Bronchial Thermoplasty With the Alair System for the Treatment of Severe Asthma
Brief Title: Research in Severe Asthma (RISA) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Narinder S Shargill, PhD., Vice President, Clinical Affairs, Asthmatx, Inc.
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Protocol #0903-27
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Results first posted 2011-11-07 (Estimated); Last update posted 2021-02-11 (Actual); Status verified 2021-01

CONDITIONS: Asthma
Keywords: Asthma; Bronchial Thermoplasty
MeSH Terms: conditions — Asthma | interventions — Bronchial Thermoplasty

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment (Experimental): Alair treatment plus standard-of-care therapy of high dose inhaled corticosteroids and long acting beta-agonists with or without oral corticosteroids at a dose of ≤ 30 mg/day.
  Interventions: Procedure: Bronchial Thermoplasty with the Alair System
- Control (Active Comparator): Standard-of-care therapy of high dose inhaled corticosteroids and long acting beta-agonists with or without oral corticosteroids at a dose of ≤30 mg/day.
  Interventions: Drug: Control

INTERVENTIONS:
Procedure: Bronchial Thermoplasty with the Alair System — Alair treatment plus standard-of-care therapy of high dose inhaled corticosteroids and long acting beta-agonists with or without oral corticosteroids at a dose of ≤ 30 mg/day.
  Other Names: Alair System
  Arms: Treatment
Drug: Control — Standard-of-care therapy of high dose inhaled corticosteroids and long acting beta-agonists with or without oral corticosteroids at a dose of ≤30 mg/day.
  Arms: Control

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of the Alair System for the treatment of severe refractory asthma.

This will be a multicenter, randomized controlled study comparing the effects of treatment with the Alair System to standard drug therapy in patients with severe asthma refractory to standard medication therapy. A total of 30 subjects will be randomized 1:1 to the Alair Group (Medical management + Alair Treatment) OR the Control Group (Medical management only).

DETAILED DESCRIPTION:
Multicenter, randomized, clinical trial conducted at 8 Investigational Sites in 3 countries.

Subjects in the Alair group to be administered the Alair treatment in 3 separate bronchoscopy sessions, while subjects in the Control group will complete 3 "Control Visits" to the Physicians office, timed to coincide with the 3 treatment bronchoscopy sessions. Following completion of all three procedures or Control Visits subjects will be evaluated at 6 weeks and 12 weeks. All subjects to remain on their maintenance asthma medications until they are evaluated again at 22 weeks after the last procedure or Control Visit. This phase from the last procedure or Control Visit out to 22 Weeks after the last procedure or Control Visit is termed the Steroid Stable Phase.

Subjects will undergo a 14 week period from 22 Weeks to 36 Weeks (termed the Steroid Wean Phase) during which an attempt will be made to wean them off either their maintenance inhaled corticosteroids (ICS) or, if taking maintenance oral corticosteroids (OCS), their oral steroids. If a subject cannot tolerate the steroid reduction at a particular level (as evidenced by loss of asthma control), they will be stabilized on their last tolerable dose of steroid.

All subjects will maintain their reduced steroid dosage from the end of the Steroid Wean Phase at 36 weeks to their final evaluations at the end of the Study at 52 weeks (termed the Reduced Steroid Phase). All subjects will be exited from the study following completion of the 52 week evaluations.

ELIGIBILITY:
Inclusion Criteria:

* Ambulatory adult; age 18-65 years
* Asthma requiring regular maintenance medication that includes high dose inhaled corticosteroid AND long acting β2 agonist (LABA) with or without other asthma maintenance medications. Oral prednisone ≤30 mg/day, leukotriene modifiers, theophylline or other asthma control drugs may be prescribed at the physician's discretion.
* Pre-bronchodilator forced expiratory volume in one second (FEV1) ≥50% predicted (patients stabilized on inhaled corticosteroids (ICS) and long acting β2 agonists)
* PC20 < 4 mg/ml per methacholine inhalation test using standardized methods, for patients with pre-bronchodilator FEV1 ≥60% predicted (or FEV1 > lower limit defined by individual hospital protocol). PC20 is the provocative concentration of Provocholine® (a brand of methacholine chloride) resulting in a drop of FEV1 of 20% or more from Baseline
* Reversible bronchoconstriction during the 12 months prior to enrollment, as demonstrated by an increase in FEV1 of at least 12% 30 minutes after 4 puffs of short-acting β2 agonist, for patients with pre-bronchodilator FEV1 < 60% predicted (or FEV1 < lower limit defined by individual hospital protocol)
* Patient must be symptomatic, despite medication with high dose inhaled corticosteroids and LABA, by at least one of the following:

  1. Use of rescue medication (short-acting β2 agonist) at least 8 of the 14 days prior to enrollment OR
  2. Daytime symptoms at least 10 of the 14 days prior to enrollment
* Non-smoker x 1 year or greater (if former smoker, less than 10 pack years total smoking history)
* Patient must be suitable for bronchoscopy in the opinion of the investigator or per hospital guidelines
* Willingness and ability to give written Informed Consent
* Willingness and ability to comply with the study protocol, including requirements for taking and abstaining from medications

Exclusion Criteria:

* Participation in another clinical trial involving respiratory intervention that could affect the outcome measures of this study, within 6 weeks prior to randomization. Patients will be disqualified from the study if they enter another study or fail to comply with prescribed asthma medications.
* Use of immunosuppressant therapy (e.g., methotrexate).
* Current or recent lower respiratory tract infection (resolved less than 6 weeks from enrollment testing)
* History of recurrent (no more than three in the last three months) lower respiratory tract infection requiring antibiotics
* Presence of other respiratory diseases including emphysema, cystic fibrosis, vocal cord dysfunction, mechanical upper airway obstruction, obstructive sleep apnea, Churg-Strauss syndrome, cardiac dysfunction, allergic bronchopulmonary aspergillosis
* DLCO (diffusion capacity) < 70% predicted
* Uncontrolled sinus disease
* Uncontrolled gastro-esophageal reflux disease
* Use of implanted electronic device such as a pacemaker or internal cardiac defibrillator
* Use of external pacemaker
* Significant co-morbid illness such as cancer, renal failure, liver disease or cerebral vascular disease
* Post-bronchodilator FEV1 of less than 55% predicted
* Known systemic hypersensitivity or contraindication to methacholine chloride or other parasympathomimetic agents
* Known sensitivity to medications required to perform bronchoscopy, including lidocaine, atropine, benzodiazepines and opioids
* Use of a systemic b-adrenergic blocking agent
* Other medical criteria.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-04; Primary Completion 2006-02 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Narinder S Shargill, PhD, Study Director — Asthmatx, Inc.

REFERENCES:
- [Derived] Pavord ID, Cox G, Thomson NC, Rubin AS, Corris PA, Niven RM, Chung KF, Laviolette M; RISA Trial Study Group. Safety and efficacy of bronchial thermoplasty in symptomatic, severe asthma. Am J Respir Crit Care Med. 2007 Dec 15;176(12):1185-91. doi: 10.1164/rccm.200704-571OC. Epub 2007 Sep 27. PMID 17901415

RESULTS

PARTICIPANT FLOW:
Groups:
- Alair: Standard-of-care therapy of high dose inhaled corticosteroids (ICS) + long acting beta agonists (LABA) ± oral corticosteroids (OCS) (≤ 30 mg/day) plus treatment with the Alair System.
- Control: Standard-of-care therapy of high dose inhaled corticosteroids (ICS) + long acting beta agonists (LABA) ± oral corticosteroids (OCS) (≤ 30 mg/day).
Period: Randomized
Arm/Group | Alair | Control
Started | 17 | 17
Completed | 15 | 17
Not Completed | 2 | 0
Period: Treatment Period
Arm/Group | Alair | Control
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0
Period: Steroid Stable (Post-Tx to 22-Weeks)
Arm/Group | Alair | Control
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0
Period: Reduced Steroid (Post-SS to 52-Weeks)
Arm/Group | Alair | Control
Started | 15 | 17
Completed | 15 | 17
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alair | Control | Total
Number analyzed (Participants) | 15 | 17 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.13 (12.97) | 42.06 (12.57) | 40.69 (12.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 7 | 16
  Male | 6 | 10 | 16
Region of Enrollment [Number; unit: participants]
  Canada | 4 | 6 | 10
  United Kingdom | 10 | 9 | 19
  Brazil | 1 | 2 | 3

OUTCOME MEASURES:

1. Primary Outcome: Respiratory Adverse Events Per Subject
Description: Respiratory adverse events (AEs) per subject reported during the Treatment Period, and Post-Treatment Period (Steroid Stable Phase, and Steroid Wean and Reduced Steroid Phase). Results were calculated by dividing the number of respiratory adverse events during each time period by the number of subjects in each group. Statistics were not calculated.
Time Frame: Baseline, 12 Months
Measure: Number; unit: Respiratory Adverse Events/Subject
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Respiratory Adverse Events/Subject
  Treatment Period | 9.1 | 3.4
  Steroid Stable Phase | 2.6 | 2.2
  Steroid Wean and Reduced Steroid Phase | 5.5 | 5.3

2. Secondary Outcome: Use of Maintenance Medications (Change From Baseline)
Description: Percent Change from Baseline at 12 Months (Steroid Wean and Reduced Steroid Phase) Follow-up Visit in dose of inhaled and/or oral corticosteroids.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Percent
  Oral Corticosteroids (OCS) | -63.5 (45.4) | -26.2 (40.7)
  Inhaled Corticosteroids (ICS) | -28.6 (30.4) | -20.0 (32.9)

3. Secondary Outcome: Use of Rescue Medications (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months (Steroid Wean and Reduced Steroid Phase) Follow-up Visits in use of rescue medications. Rescue medications for asthma are short-acting beta-agonists that bring quick relief of asthma symptoms.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Puffs/7 Days
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Puffs/7 Days
  Steroid Stable Phase | -26.56 (40.05) | -1.47 (11.66)
  Steroid Wean and Reduced Steroid Phase | -25.56 (31.19) | -6.07 (12.43)

4. Secondary Outcome: Total Symptom Score (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months (Steroid Wean and Reduced Steroid Phase) Follow-up Visits in Total Symptom Score. The Total Symptom Score comprises the sum of six asthma symptom measurements recorded in a Daily Diary. Each of these symptoms is scored on a scale of 0 to 3 each day by the subject. The sum of the scores for these 6 symptoms comprises the Total Symptom Score, which measures overall asthma symptoms. The maximum score possible is 18. A lower Total Symptom Score represents better asthma control.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Units on a scale
  Steroid Stable Phase | -1.75 (2.58) | -0.89 (1.84)
  Steroid Wean and Reduced Steroid Phase | -1.37 (2.61) | -1.21 (1.63)

5. Secondary Outcome: Pre-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months (Steroid Wean and Reduced Steroid Phase) Follow-up Visits in forced expiratory volume in one second (FEV1). FEV1 is the volume of air expired during the first second of a maximal effort expiration started at total lung capacity.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Percent Change
  Steroid Stable Phase | 14.91 (17.40) | -0.94 (22.34)
  Steroid Wean and Reduced Steroid Phase | 7.97 (19.13) | 1.89 (15.00)

6. Secondary Outcome: Post-Bronchodilator FEV1 (Percent Predicted) (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months(Steroid Wean and Reduced Steroid Phase) Follow-up Visits in forced expiratory volume in one second (FEV1). FEV1 is the volume of air expired during the first second of a maximal effort expiration started at total lung capacity.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Percent Change
  Steroid Stable Phase | 5.74 (8.56) | -0.82 (16.78)
  Steroid Wean and Reduced Steroid Phase | 2.76 (11.57) | -1.90 (11.97)

7. Secondary Outcome: Asthma Control Questionnaire (ACQ) Score (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months (Steroid Wean and Reduced Steroid Phase) Follow-up Visits in Asthma Control Questionnaire (ACQ) score. The ACQ is a self-administered patient questionnaire that assesses individual subject asthma control. The ACQ comprises 6 questions that relate to the patient's asthma symptoms, activity limitations, and daily rescue bronchodilator use, and FEV1. Each question is scored from 0 (Better) to 6 (Worse). The ACQ is based on a one-week recall period. A decrease in the ACQ score indicates better asthma control.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Units on a scale
  Steroid Stable Phase | -1.04 (1.03) | -0.13 (1.00)
  Steroid Wean and Reduced Steroid Phase | -0.99 (0.83) | -0.22 (0.78)

8. Secondary Outcome: Asthma Quality of Life Questionnaire (AQLQ) Score (Change From Baseline)
Description: Change from Baseline at 22-Weeks (Steroid Stable Phase) and 12 Months(Steroid Wean and Reduced Steroid Phase) Follow-up Visits in Asthma Quality of Life Questionnaire (AQLQ) score. The AQLQ is a self-administered patient questionnaire that assesses four aspects or domains of daily life for patients with asthma: symptoms, emotional function, activity limitations, and environmental stimuli. The AQLQ is based on a 2-week recall period and consists of 32 questions, each scored from 1 (Worse) to 7 (Better). An increase in the AQLQ score indicates a better quality of life.
Time Frame: Baseline, 12 Months
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Alair | Control
Number analyzed (Participants) | 15 | 17
Units on a scale
  Steroid Stable Phase | 1.21 (1.05) | 0.15 (0.75)
  Steroid Wean and Reduced Steroid Phase | 1.53 (0.79) | 0.42 (0.82)

ADVERSE EVENTS:
Arm/Group | Alair (Treatment Period) | Control (Treatment Period) | Alair (Steroid Stable Phase) | Control (Steroid Stable Phase) | Alair (Steroid Wean and Reduced Steroid Phases) | Control (Steroid Wean and Reduced Steroid Phases)
Serious Adverse Events (participants affected / at risk) | 5/15 | 1/17 | 4/15 | 1/17 | 2/15 | 1/17
Other Adverse Events (participants affected / at risk) | 15/15 | 17/17 | 15/15 | 15/17 | 15/15 | 15/17
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=15) | Control (Treatment Period) (N=17) | Alair (Steroid Stable Phase) (N=15) | Control (Steroid Stable Phase) (N=17) | Alair (Steroid Wean and Reduced Steroid Phases) (N=15) | Control (Steroid Wean and Reduced Steroid Phases) (N=17)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 0 | 0 | 1
Dyspnoea/Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 2 | 1
Gallbladder Pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0
Hernia Repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alair (Treatment Period) (N=15) | Control (Treatment Period) (N=17) | Alair (Steroid Stable Phase) (N=15) | Control (Steroid Stable Phase) (N=17) | Alair (Steroid Wean and Reduced Steroid Phases) (N=15) | Control (Steroid Wean and Reduced Steroid Phases) (N=17)
Abdominal Discomfort (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 4 | 0 | 1 | 0 | 1 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1 | 1
Anaesthetic Complication (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 0 | 1 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Arthropod Sting (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Arthroscopic Surgery (Surgical and medical procedures) | 0 | 0 | 0 | 0 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 0 | 0
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 3 | 1 | 2
Breast Mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Breath Sounds Decreased (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Bronchial Irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0 | 0 | 0 | 0
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chapped Lips (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Chest Discomfort (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 1 | 2 | 2 | 6
Chest Pain (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 0 | 1 | 1
Chest Wall Pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 4 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11 | 6 | 2 | 4 | 6 | 4
Crackles Lung (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Dandruff (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dermatitis Allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 4 | 2 | 1 | 1 | 2
Difficulty In Walking (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 4 | 0 | 0 | 0 | 1 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 9 | 5 | 5 | 7 | 8 | 10
Dyspnoea Exacerbated (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2 | 0 | 1 | 4
Ear Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 0
Eye Inflammation (Eye disorders) | 0 | 1 | 0 | 0 | 0 | 0
Eye Pruritis (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 3 | 1 | 0
Gallbladder Pain (Hepatobiliary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Gastroesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Headache (Nervous system disorders) | 3 | 4 | 1 | 3 | 4 | 2
Hernia Repair (Surgical and medical procedures) | 0 | 1 | 0 | 0 | 0 | 0
Herpes Simplex (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 0
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Infected Insect Bite (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 2 | 0 | 1 | 0 | 0 | 0
Influenza Like Illness (General disorders) | 0 | 1 | 0 | 1 | 0 | 1
Infusion Site Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 1 | 0 | 1 | 1 | 0
Irritability (Psychiatric disorders) | 0 | 1 | 0 | 0 | 0 | 0
Joint Injury (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0 | 0 | 0
Joint Swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 2 | 0
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0
Limb Injury (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 1 | 0
Localised Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Localised Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Lower Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 2 | 5 | 2 | 2 | 6 | 2
Meniscus Lesion (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Muscle Cramp (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 1
Musculoskeletal Chest Pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Musculoskeletal Stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Nail Operation (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 2 | 1 | 3 | 4
Nasopharyngitis (Infections and infestations) | 3 | 3 | 2 | 1 | 4 | 4
Nausea (Gastrointestinal disorders) | 4 | 1 | 1 | 1 | 0 | 2
Neuropathic Pain (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Nocturnal Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 3 | 0 | 0 | 0
Oedema (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Oedema Peripheral (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Oral Candidiasis (Infections and infestations) | 2 | 1 | 3 | 0 | 0 | 1
Otitis Media (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1 | 0
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 1 | 1 | 0 | 0 | 2 | 0
Pancreatic Cyst (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Pharyngolaryngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 1 | 2 | 0
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Post Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 8 | 4 | 2 | 4 | 8 | 1
Pyrexia (General disorders) | 1 | 2 | 1 | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rectal Haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 2 | 1
Sinus Headache (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Skin Chapped (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Skin Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1 | 0
Sputum Discoloured (Respiratory, thoracic and mediastinal disorders) | 6 | 2 | 0 | 2 | 3 | 4
Stomach Discomfort (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Subcutaneous Abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0
Thirst (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Thyroid Pain (Endocrine disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tooth Abscess (Infections and infestations) | 1 | 0 | 0 | 0 | 1 | 0
Tooth Extraction (Surgical and medical procedures) | 0 | 0 | 1 | 0 | 0 | 0
Tooth Fracture (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Tooth Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Tremor (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 3 | 1 | 6 | 4
Urinary Tract Infection (Infections and infestations) | 2 | 1 | 1 | 0 | 0 | 1
Vaginal Candidiasis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Vaginal Infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 3 | 3 | 1 | 0 | 2 | 0
Weight Increased (Investigations) | 1 | 0 | 0 | 0 | 0 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 11 | 4 | 6 | 2 | 5 | 10
Wound Infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less